CLINICAL TRIAL: NCT03060629
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2b Efficacy Study of a Heterologous Prime/Boost Vaccine Regimen of Ad26.Mos4.HIV and Aluminum Phosphate-adjuvanted Clade C gp140 in Preventing HIV-1 Infection in Adult Women in Sub-Saharan Africa
Brief Title: A Study to Assess the Efficacy of a Heterologous Prime/Boost Vaccine Regimen of Ad26.Mos4.HIV and Aluminum Phosphate-Adjuvanted Clade C gp140 in Preventing Human Immunodeficiency Virus (HIV) -1 Infection in Women in Sub-Saharan Africa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by the sponsor after the last participant completed the Month 24 visit as the pre-specified criteria to continue the study were not met.
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108263; VAC89220HPX2008 (Other: Janssen Vaccines & Prevention B.V.); HVTN 705 (Other: Janssen Vaccines & Prevention B.V.); HVTN 705/VAC89220HPX2008 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: HIV-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor will be also blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will receive Ad26.Mos4.HIV 5*10^10 virus particles (vp) as 0.5 milliliter (mL) via Intramuscular (IM) injection into the left deltoid on Months 0, 3, 6, and 12 and Clade C gp140 (250 [microgram] mcg) mixed with Aluminum phosphate adjuvant as 0.5 mL IM into the right deltoid on Months 6 and 12.
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C gp140
- Group 2 (Placebo Comparator): Participants will receive Placebo for Ad26.Mos4.HIV as 0.5 mL into the left deltoid on Months 0, 3, 6, and 12 and Placebo for Clade C gp140 / Aluminum phosphate adjuvant as 0.5 mL IM into the right deltoid on Months 6 and 12.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.Mos4.HIV — Participants will receive Ad26.Mos4.HIV 5x10^10 virus particles (vp) as 0.5 milliliter (mL) via Intramuscular (IM) into the left deltoid on Months 0, 3, 6, and 12.
  Arms: Group 1
Biological: Clade C gp140 — Participants will receive Clade C gp140 (250 mcg) mixed with Aluminum phosphate adjuvant as 0.5 mL IM into the right deltoid on Months 6 and 12.
  Arms: Group 1
Biological: Placebo — Participants will receive matching placebo.
  Arms: Group 2

SUMMARY:
The primary purpose of this study is to assess the preventive vaccine efficacy (VE), safety and tolerability of a heterologous prime/boost regimen utilizing Ad26.Mos4.HIV and aluminum-phosphate adjuvanted Clade C gp 140 for the prevention of Human Immuno Virus (HIV) infection in HIV-seronegative women residing in sub-Saharan Africa from confirmed HIV-1 infections diagnosed between the Month 7 and Month 24 visits.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active, defined as having had sexual intercourse with a male partner at least twice in the past 30 days prior to screening, and is considered by the site staff to be at risk for Human Immunodeficiency Virus (HIV) infection
* Access to a participating HIV Vaccine Trials Network (HVTN) Clinical Research Sites (CRS) and willingness to be followed for the planned duration of the study
* Willingness to discuss HIV infection risks and willing to receive HIV risk reduction counseling and appropriate referrals to minimize HIV acquisition, as applicable
* Negative beta human chorionic gonadotropin (beta-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing
* Participants must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until 3 months after the last vaccination

Exclusion Criteria:

* Investigational research agents received within 30 days before first vaccination
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 705/HPX2008 (Protocol Safety Review Team) PSRT will determine eligibility on a case-by-case basis
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (example: measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (example, tetanus, pneumococcal, Hepatitis A or B)
* Immunosuppressive medications received within 6 months before first vaccination

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2636 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (23):
- UNC Lilongwe Project, Lilongwe, Malawi
- Polana Caniço Health Research and Training Center (CISPOC), Maputo, Mozambique
- South Africa (16):
  - Josha Research, Bloemfontein
  - Masiphumelele Research Centre, Cape Town
  - Ndlovu Elandsdoorn Site, Dennilton
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Diepkloof
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Johannesburg
  - The Aurum Institute Klerksdorp Clinical Research Centre, Klerksdorp
  - Qhakaza Mbokodo Research Centre, KwaZulu-Natal
  - South African Medical Research Council Chatsworth Clinical Research Site, KwaZulu-Natal
  - Centre for the AIDS Programme of Research in South Africa, KwaZulu-Natal
  - South African Medical Research Council Tongaat Clinical Research Site, KwaZulu-Natal
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - Nelson Mandela Academic Clinical Research Unit 'NeMACRU', Mthatha
  - MeCRU Clinical Research Unit, Pretoria
  - The Aurum Institute Rustenburg Clinical Research Site, Rustenburg
  - Setshaba Research Centre, Soshanguve
  - The Aurum Institute: Tembisa - Clinic 4, Tembisa
- Zambia (3):
  - Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka
  - Center for Family Health Research in Zambia (CFHRZ), Lusaka
  - Center for Family Health Research in Zambia (CFHRZ), Ndola
- Zimbabwe (2):
  - St Mary's Clinic, Chitungwiza
  - University of Zimbabwe-UCSF, Harare - Seke South

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Gray GE, Mngadi K, Lavreys L, Nijs S, Gilbert PB, Hural J, Hyrien O, Juraska M, Luedtke A, Mann P, McElrath MJ, Odhiambo JA, Stieh DJ, van Duijn J, Takalani AN, Willems W, Tapley A, Tomaras GD, Van Hoof J, Schuitemaker H, Swann E, Barouch DH, Kublin JG, Corey L, Pau MG, Buchbinder S, Tomaka F; Imbokodo/HVTN 705/HPX2008 Study Group. Mosaic HIV-1 vaccine regimen in southern African women (Imbokodo/HVTN 705/HPX2008): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Infect Dis. 2024 Nov;24(11):1201-1212. doi: 10.1016/S1473-3099(24)00358-X. Epub 2024 Jul 19. PMID 39038477
- [Derived] Barouch DH, Tomaka FL, Wegmann F, Stieh DJ, Alter G, Robb ML, Michael NL, Peter L, Nkolola JP, Borducchi EN, Chandrashekar A, Jetton D, Stephenson KE, Li W, Korber B, Tomaras GD, Montefiori DC, Gray G, Frahm N, McElrath MJ, Baden L, Johnson J, Hutter J, Swann E, Karita E, Kibuuka H, Mpendo J, Garrett N, Mngadi K, Chinyenze K, Priddy F, Lazarus E, Laher F, Nitayapan S, Pitisuttithum P, Bart S, Campbell T, Feldman R, Lucksinger G, Borremans C, Callewaert K, Roten R, Sadoff J, Scheppler L, Weijtens M, Feddes-de Boer K, van Manen D, Vreugdenhil J, Zahn R, Lavreys L, Nijs S, Tolboom J, Hendriks J, Euler Z, Pau MG, Schuitemaker H. Evaluation of a mosaic HIV-1 vaccine in a multicentre, randomised, double-blind, placebo-controlled, phase 1/2a clinical trial (APPROACH) and in rhesus monkeys (NHP 13-19). Lancet. 2018 Jul 21;392(10143):232-243. doi: 10.1016/S0140-6736(18)31364-3. Epub 2018 Jul 6. PMID 30047376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For Participant Flow below, data were summarized based on assigned treatment.
Groups:
- Group 1: Ad26.Mos.HIV Vaccine: Participants received adenovirus serotype 26-Mosaic-Human Immunodeficiency Virus (Ad26.Mos4.HIV) 5*10^10 virus particles (vp) per 0.5 milliliter (mL) via Intramuscular (IM) injection at Months 0, 3, 6, and 12 and Clade C glycoprotein (gp) 140 (250 [micrograms] mcg) mixed with aluminum phosphate adjuvant 425 mcg per 0.5 mL IM injection at Months 6 and 12.
- Group 2: Placebo: Participants received Placebo matching to Ad26.Mos4.HIV as 0.5 mL via IM injection at Months 0, 3, 6, and 12 and Placebo matching to Clade C gp140/aluminum phosphate adjuvant as 0.5 mL IM injection at Months 6 and 12.
Period: Overall Study
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Started | 1313 | 1323
Completed | 78 | 88
Not Completed | 1235 | 1235
Not completed — Death | 4 | 5
Not completed — Withdrawal by Subject | 50 | 35
Not completed — Unable to Adhere to Visit Schedule | 21 | 23
Not completed — Participant Relocate | 15 | 15
Not completed — Unable to Contact Participant | 34 | 23
Not completed — Investigator Decision | 7 | 7
Not completed — Study Terminated by Sponsor | 1100 | 1123
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo | Total
Number analyzed (Participants) | 1313 | 1323 | 2636
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [18 to 35] | 23 [18 to 35] | 23 [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1313 | 1323 | 2636
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1313 | 1323 | 2636
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1302 | 1317 | 2619
  Colored/Mixed | 5 | 4 | 9
  Indian | 2 | 0 | 2
  Multiple | 1 | 0 | 1
  White | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  MALAWI | 78 | 79 | 157
  MOZAMBIQUE | 23 | 22 | 45
  SOUTH AFRICA | 882 | 892 | 1774
  ZAMBIA | 164 | 165 | 329
  ZIMBABWE | 166 | 165 | 331

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Immuno Deficiency Virus-1 (HIV-1) Infection Diagnosed Between Month 7 to Month 24 Post Enrollment
Description: Number of participants with HIV-1 infection diagnosed between Month 7 to Month 24 post enrollment was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: Month 7 up to Month 24
Population: Per protocol (PP) population set included participants from the full analysis set (FAS; all randomized participants who received at least one study vaccine administration) who were HIV-1 uninfected 4 weeks after the third vaccination visit, who received all planned vaccinations at the first 3 vaccination visits within the respective visit windows and had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1080 | 1108
Participants | 54 | 65

2. Primary Outcome: Percentage of Participants With Local Reactogenicity Signs and Symptoms After First Vaccination
Description: Percentage of participants with local reactogenicity signs and symptoms after first vaccination were reported. Local reactogenicity events (solicited local adverse events) were defined as events at the injection site. Local reactogenicity signs and symptoms included pain and/or tenderness proximal to the injection site.
Time Frame: Up to 7 days after first vaccination on Day 0 (Day 7)
Population: FAS included all randomized participants who received at least 1 vaccine administration. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. The safety analyses were performed based on the actual treatment that the participants received after the first vaccination. Hence, one participant from Group 2 was analyzed in Group 1 for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1316 | 1320
Percentage of participants | 34.2 | 9.4

3. Primary Outcome: Percentage of Participants With Local Reactogenicity Signs and Symptoms After Second Vaccination
Description: Percentage of participants with local reactogenicity signs and symptoms after second vaccination was reported. Local reactogenicity events (solicited local adverse events) were defined as events at the injection site. Local reactogenicity signs and symptoms included pain and/or tenderness proximal to the injection site.
Time Frame: Up to 7 days after second vaccination on Day 84 (Day 91)
Population: FAS included all randomized participants who received at least 1 vaccine administration. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1190 | 1215
Percentage of participants | 20.0 | 8.1

4. Primary Outcome: Percentage of Participants With Local Reactogenicity Signs and Symptoms After Third Vaccination
Description: Percentage of participants with local reactogenicity signs and symptoms after third vaccination was reported. Local reactogenicity events (solicited local adverse events) were defined as events at the injection site. Local reactogenicity signs and symptoms included pain and/or tenderness proximal to the injection site.
Time Frame: Up to 7 days after third vaccination on Day 168 (Up to Day 175)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1160 | 1188
Percentage of participants | 25.2 | 8.9

5. Primary Outcome: Percentage of Participants With Local Reactogenicity Signs and Symptoms After Fourth Vaccination
Description: Percentage of participants with local reactogenicity signs and symptoms after fourth vaccination was reported. Local reactogenicity events (solicited local adverse events) were defined as events at the injection site. Local reactogenicity signs and symptoms included pain and/or tenderness proximal to the injection site.
Time Frame: Up to 7 days after fourth vaccination on Day 364 (Up to Day 371)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1099 | 1111
Percentage of participants | 25.7 | 8.6

6. Primary Outcome: Percentage of Participants With Systematic Reactogenicity Signs and Symptoms After First Vaccination
Description: Percentage of participants with systematic reactogenicity signs and symptoms after first vaccination was reported. Systemic reactogenicity events (solicited systemic adverse events) defined as events occurred in a predefined post-vaccination period for which the subject was specifically questioned. Systemic reactogenicity signs and symptoms included increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting.
Time Frame: Up to 7 days after first vaccination on Day 0 (Day 7)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1316 | 1320
Percentage of participants | 52.9 | 40.9

7. Primary Outcome: Percentage of Participants With Systematic Reactogenicity Signs and Symptoms After Second Vaccination
Description: Percentage of participants with systematic reactogenicity signs and symptoms after second vaccination was reported. Systemic reactogenicity events (solicited systemic adverse events) defined as events occurred in a predefined post-vaccination period for which the subject was specifically questioned. Systemic reactogenicity signs and symptoms included increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting.
Time Frame: Up to 7 days after second vaccination on Day 84 (Day 91)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1190 | 1215
Percentage of participants | 33.2 | 28.6

8. Primary Outcome: Percentage of Participants With Systematic Reactogenicity Signs and Symptoms After Third Vaccination
Description: Percentage of participants with systematic reactogenicity signs and symptoms after third vaccination was reported. Systemic reactogenicity events (solicited systemic adverse events) defined as events occurred in a predefined post-vaccination period for which the subject was specifically questioned. Systemic reactogenicity signs and symptoms included increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting.
Time Frame: Up to 7 days after third vaccination on Day 168 (Up to Day 175)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1160 | 1188
Percentage of participants | 31.5 | 26.8

9. Primary Outcome: Percentage of Participants With Systematic Reactogenicity Signs and Symptoms After Fourth Vaccination
Description: Percentage of participants with systematic reactogenicity signs and symptoms after fourth vaccination was reported. Systemic reactogenicity events (solicited systemic adverse events) defined as events occurred in a predefined post-vaccination period for which the subject was specifically questioned. Systemic reactogenicity signs and symptoms included increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting.
Time Frame: Up to 7 days after fourth vaccination on Day 364 (Up to Day 371)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1099 | 1111
Percentage of participants | 29.4 | 23.6

10. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs) for 30 Days After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a study product and which does not necessarily have a causal relationship with the study treatment. The most frequent unsolicited AEs were upper respiratory tract infection, back pain, cough, and hypertension.
Time Frame: 30 days after first vaccination on Day 0 (Up to Day 30)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1316 | 1320
Percentage of participants | 16.6 | 14.8

11. Primary Outcome: Percentage of Participants With Unsolicited AEs for 30 Days After Second Vaccination
Description: as for outcome 10
Time Frame: 30 days after second vaccination on Day 84 (Up to Day 114)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1190 | 1215
Percentage of participants | 17.1 | 15.1

12. Primary Outcome: Percentage of Participants With Unsolicited AEs for 30 Days After Third Vaccination
Description: as for outcome 10
Time Frame: 30 days after third vaccination on Day 168 (Up to Day 198)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1160 | 1188
Percentage of participants | 39.8 | 40.3

13. Primary Outcome: Percentage of Participants With Unsolicited AEs for 30 Days After Fourth Vaccination
Description: as for outcome 10
Time Frame: 30 days after fourth vaccination on Day 364 (Up to Day 394)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1099 | 1111
Percentage of participants | 63.5 | 62.5

14. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a study product and which does not necessarily have a causal relationship with the study treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to Month 36 (up to end of the study)
Population: FAS included all randomized participants who received at least 1 vaccine administration. The safety analyses were performed based on the actual treatment that the participants received.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1317 | 1319
Percentage of participants | 3.7 | 2.8

15. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: Percentage of participants with AESIs was reported. Immune-mediated diseases were considered as AESIs in this study.
Time Frame: Up to Month 36 (up to end of the study)
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1317 | 1319
Percentage of participants | 0.2 | 0.2

16. Primary Outcome: Percentage of Participants With AEs Leading to Early Participant Withdrawal or Early Discontinuation of Study Product
Description: Percentage of participants with AEs leading to early participant withdrawal or early discontinuation of study product were reported. An AE is any untoward medical occurrence in a clinical investigation participant administered a study product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to Month 36 (up to end of the study)
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1317 | 1319
Percentage of participants | 0.2 | 0.2

17. Secondary Outcome: Number of Participants With HIV-1 Infection Diagnosed From Enrollment (Baseline) Through Month 24 Post Enrollment
Description: Number of participants with HIV-1 infection diagnosed from enrollment (baseline) through month 24 post enrollment was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: Baseline up to Month 24
Population: Modified Intent-to-Treat (MITT) analysis set included participants in the FAS who were HIV-1 uninfected on the date of first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1311 | 1319
Participants | 91 | 102

18. Secondary Outcome: Number of Participants With HIV-1 Infection Diagnosed From Enrollment (Baseline) Through Month 36 (End of Study) Post Enrollment
Description: Number of participants with HIV-1 infection diagnosed from enrollment (baseline) through Month 36 post enrollment was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: Baseline up to Month 36 (End of study)
Population: MITT analysis set included participants in the FAS who were HIV-1 uninfected on the date of first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1311 | 1319
Participants | 115 | 127

19. Secondary Outcome: Number of Participants With HIV-1 Infection Diagnosed From Month 13 Through Month 24 Post Enrollment
Description: Number of participants with HIV-1 infection diagnosed from Month 13 through Month 24 post enrollment was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: Month 13 up to Month 24
Population: Full immunization set (FIS) included participants in the FAS who were HIV-1 uninfected 4 week after the fourth vaccination visit and who received all planned vaccinations within the respective visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 981 | 995
Participants | 32 | 35

20. Secondary Outcome: Number of Participants With HIV-1 Infection Diagnosed From Month 13 Through Month 36 (End of Study) Post Enrollment
Description: Number of participants with HIV-1 infection diagnosed from Month 13 through Month 36 (end of study) post enrollment was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: Month 13 up to Month 36 (End of study)
Population: FIS included participants in the FAS who were HIV-1 uninfected 4 week after the fourth vaccination visit and who received all planned vaccinations within the respective visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 981 | 995
Participants | 53 | 58

21. Secondary Outcome: Geometric Mean of Binding Antibody Responses to HIV Envelop (ENV) Clade (gp140) C (ZA) Analyzed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: A weighted geometric mean of the binding antibody responses to HIV envelope (ENV) gp140 Clade C 97ZA protein analyzed by ELISA was reported.
Time Frame: Months 0, 7, 13 and 24
Population: FIS included participants in the FAS who were HIV-1 uninfected 4 weeks after the fourth vaccination visit and who received all planned vaccinations within the respective visit windows. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 50 | 10
ELISA Units per milliliter (EU/mL)
  Month 0 | 53 [45 to 63] | 43 [37 to 49]
  Month 7 | 38834 [26484 to 56942] | 43 [37 to 49]
  Month 13 | 66147 [50523 to 86602] | 62 [36 to 109]
  Month 24 | 5920 [4559 to 7688] | 49 [33 to 72]

22. Secondary Outcome: Geometric Mean of Interferon-gamma (IFN-gamma) T-Cells Responses Analyzed by Enzyme-linked Immunospot Assay (ELISpot)
Description: Geometric mean of IFN-gamma T-cells responses analyzed by ELISpot were reported. A weighted geometric mean of the number of spot-forming cells (SFC) per million peripheral blood mononuclear cells (PBMCs) producing Interferon-gamma upon stimulation with potential T-cell epitope (PTE) ENV peptide pools analyzed by ELISpot was reported. Reported responses are the sum of the number of SFCs/10^6 PBMCS for PTE Env1, Env2 and Env3 sub-pools.
Time Frame: Months 0, 7, 13 and 24
Population: FIS included participants who were HIV-1 uninfected 4 week after the fourth vaccination visit and who received all planned vaccinations within the respective visit windows. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/million PBMCs
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 50 | 10
SFC/million PBMCs
  Month 0 | 33.5 [29.7 to 33.7] | 30.0 [30.0 to 30.0]
  Month 7: number analyzed (Participants) | 50 | 9
  Month 7 | 241.2 [168.0 to 346.2] | 33.9 [26.7 to 43.0]
  Month 13: number analyzed (Participants) | 49 | 10
  Month 13 | 287.1 [201.3 to 409.5] | 33.2 [28.8 to 38.2]
  Month 24: number analyzed (Participants) | 50 | 9
  Month 24 | 172.7 [117.0 to 254.8] | 30.8 [29.2 to 32.5]

23. Secondary Outcome: Number of Participants With Viral Sequences
Description: Number of participants with viral sequences were reported. Viral sequencing was conducted on the earliest available plasma specimens with positive HIV-1 ribose nucleic acid polymerase chain reaction (RNA PCR) tests from study participants who were diagnosed with HIV-1 infection.
Time Frame: Month 7 up to Month 24
Population: PP population set included participants from the FAS; all randomized participants who received at least one study vaccine administration) who were HIV-1 uninfected 4 weeks after the third vaccination visit, who received all planned vaccinations at the first 3 vaccination visits within the respective visit windows and had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
Number analyzed (Participants) | 1080 | 1108
Participants | 51 | 63

ADVERSE EVENTS:
Time Frame: Up to Month 36
Description: Full analysis set (FAS) included all randomized participants who received at least 1 vaccine administration. Here, N (total number of participants at risk) signifies participants who were assessed for AEs as safety analyses were performed based on the actual treatment that the participants received. Therefore, number of participants affected for all-cause mortality are different in participant flow section and adverse event section.
Arm/Group | Group 1: Ad26.Mos.HIV Vaccine | Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 5/1317 | 4/1319
Serious Adverse Events (participants affected / at risk) | 49/1317 | 37/1319
Other Adverse Events (participants affected / at risk) | 798/1317 | 806/1319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26.Mos.HIV Vaccine (N=1317) | Group 2: Placebo (N=1319)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 2 | 2
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1
Gonococcal pelvic inflammatory disease (Infections and infestations) | 0 | 1
HIV-associated neurocognitive disorder (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Wound sepsis (Infections and infestations) | 1 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 2 | 0
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 1 | 0
Psychogenic seizure (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 4 | 2
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Maternal death during childbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcoholic psychosis (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 2
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26.Mos.HIV Vaccine (N=1317) | Group 2: Placebo (N=1319)
Genitourinary chlamydia infection (Infections and infestations) | 528 | 527
Genitourinary tract gonococcal infection (Infections and infestations) | 269 | 288
Syphilis (Infections and infestations) | 69 | 79
Upper respiratory tract infection (Infections and infestations) | 79 | 77
Vulvovaginitis trichomonal (Infections and infestations) | 245 | 239
Vaginal discharge (Reproductive system and breast disorders) | 102 | 113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03060629/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT03060629/SAP_001.pdf